CLINICAL TRIAL: NCT03371225
Title: Optimized tDCS for Fibromyalgia: Targeting the Endogenous Pain Control System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Felipe Fregni, MD, PhD, MPH, Director of Spaulding Neuromodulation Center, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Other
Other Study IDs: 2017P002524
Record Dates: First submitted 2017-11-20; First posted 2017-12-13 (Actual); Results first posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Transcranial Direct Current Stimulation; Muscle Stretching Exercises; Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (4):
- Active tDCS and Active Exercise (Experimental): Active tDCS for 20 min Active exercise (60-70% max HR) for 30 min
  Interventions: Device: Active tDCS; Procedure: Active Exercise
- Sham tDCS and Active Exercise (Active Comparator): Sham tDCS for 20 min Active exercise (60-70% max HR) for 30 min
  Interventions: Procedure: Active Exercise; Device: Sham tDCS
- Active tDCS and Sham Exercise (Active Comparator): Active tDCS for 20 min Sham exercise (within 10% baseline HR) for 30 min
  Interventions: Device: Active tDCS; Procedure: Sham Exercise
- Sham TDCS and Sham Exercise (Sham Comparator): Sham tDCS for 20 min Sham exercise (within 10% baseline HR) for 30 min
  Interventions: Device: Sham tDCS; Procedure: Sham Exercise

INTERVENTIONS:
Device: Active tDCS — Active tDCS: A 1x1 Low-intensity DC Stimulator will be used to deliver direct current through rubber electrodes in saline soaked sponges. The anode will be placed over the left primary motor cortex (M1) while the cathode will be placed over the contralateral supra-orbital area. 20 minutes of tDCS will be applied.
  Other Names: tDCS
  Arms: Active tDCS and Active Exercise; Active tDCS and Sham Exercise
Procedure: Active Exercise — Participants will walk briskly in a treadmill (as to keep at 60-70% maximum heart rate) for 30 minutes
  Other Names: Aerobic Exercises
  Arms: Active tDCS and Active Exercise; Sham tDCS and Active Exercise
Device: Sham tDCS — Active tDCS: A 1x1 Low-intensity DC Stimulator will be used to deliver direct current through rubber electrodes in saline soaked sponges. The anode will be placed over the left primary motor cortex (M1) while the cathode will be placed over the contralateral supra-orbital area. Only 30 seconds of current will be applied for the sham condition.
  Other Names: Placebo tDCS
  Arms: Sham TDCS and Sham Exercise; Sham tDCS and Active Exercise
Procedure: Sham Exercise — Participants will walk in a treadmill (as to keep at 10% within their baseline heart rate) for 30 minutes.
  Other Names: Placebo Aerobic Exercise
  Arms: Active tDCS and Sham Exercise; Sham TDCS and Sham Exercise

SUMMARY:
This trial aims at understanding the mechanisms of optimized transcranial direct current stimulation (tDCS) (16 tDCS sessions combined with exercise)] on pain control. Optimized tDCS can lead to stronger engagement of the endogenous pain regulatory system that will ultimately lead to increased pain relief in patients with fibromyalgia (FM). Therefore, the investigators designed a 2x2 factorial mechanistic trial [tDCS (active and sham) and aerobic exercise (AE) (active and control)] to evaluate the effects of 4 weeks of tDCS coupled with exercise on the endogenous pain regulatory system assessed by conditioned pain modulation (CPM) and central sensitization as assessed by temporal slow pain summation (TSPS), and compared to either intervention alone and to no intervention.

DETAILED DESCRIPTION:
Recent evidence has suggested that FM pain can be related to deficits in pain endogenous regulatory control and that novel non-pharmacological interventions, such as tDCS can modulate this system and, consequently, reduce pain intensity. Widespread pain in FM is thought to represent enhanced pain sensitivity that is maintained by central mechanisms. This suggests changes in the descending pain control mechanisms and a possible relationship with the central sensitization phenomenon. Recent evidence has suggested that pain inhibitory pathways are affected in FM; thus, further understanding these pathways' role can significantly change how the treatment of this condition. In this study the investigators will test the effects of two interventions -tDCS and aerobic exercise - on the modulation of the endogenous inhibitory pain system in fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

1. Age range 18-65 years,
2. Diagnosis of FM pain according to the ACR 2010 criteria (existing pain for more than 6 months with an average of at least 4 on a 0-10 VAS scale) without other comorbid chronic pain diagnosis,
3. Pain resistant to common analgesics and medications for chronic pain such as Tylenol, Aspirin, Ibuprofen, Soma, Parafon Forte DCS, Zanaflex, and Codeine,
4. Must have the ability to feel sensation by Von-Frey fiber on the forearm,
5. Able to provide informed consent to participate in the study.

Exclusion Criteria:

1. Clinically significant or unstable medical or psychiatric disorder,
2. history of substance abuse within the past 6 months as self-reported (if subject reports a history of substance abuse, we will confirm using DSM V criteria),
3. Previous significant neurological history (e.g., traumatic brain injury), resulting in neurological deficits, such as cognitive or motor deficits, as self-reported,
4. Previous neurosurgical procedure with craniotomy,
5. Severe depression (If a patient scores >30 on the Beck Depression Inventory, one will obtain clearance. If one does not pass the medical clearance, one will not be included in the study)
6. Pregnancy (as the safety of tDCS in pregnant population (and children) has not been assessed (though risk is non-significant), the investigators will exclude pregnant women (and children). Women of child-bearing potential will be required to take a urine pregnancy test during the screening process and at every week of stimulation),
7. Current opiate use in large doses (more than 30mg of oxycodone/hydrocodone or 7.5mg of hydromorphone (Dilaudid) or equivalent),
8. Patients will be excluded when they have increased risk for exercise

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2024-09-26 (Actual); Study Completion 2025-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Fregni, MD PhD MPH, Principal Investigator — Spaulding Rehabilitation Hospital
Locations (1):
- Spaulding Rehabilitation Hospital for Continuing Care, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon completion of the trial and after publication of the primary manuscript, we plan to publish the de-identified dataset following the guidelines of our institution (Spaulding Rehabilitation Hospital/Partners Healthcare and Harvard Medical School).

REFERENCES:
- [Derived] Pacheco-Barrios K, Teixeira PEP, Martinez-Magallanes D, Neto MS, Pichardo EA, Camargo L, Lima D, Cardenas-Rojas A, Fregni F. Brain compensatory mechanisms in depression and memory complaints in fibromyalgia: the role of theta oscillatory activity. Pain Med. 2024 Aug 1;25(8):514-522. doi: 10.1093/pm/pnae030. PMID 38652585
- [Derived] Castelo-Branco L, Uygur Kucukseymen E, Duarte D, El-Hagrassy MM, Bonin Pinto C, Gunduz ME, Cardenas-Rojas A, Pacheco-Barrios K, Yang Y, Gonzalez-Mego P, Estudillo-Guerra A, Candido-Santos L, Mesia-Toledo I, Rafferty H, Caumo W, Fregni F. Optimised transcranial direct current stimulation (tDCS) for fibromyalgia-targeting the endogenous pain control system: a randomised, double-blind, factorial clinical trial protocol. BMJ Open. 2019 Oct 30;9(10):e032710. doi: 10.1136/bmjopen-2019-032710. PMID 31672712

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 116 subjects were enrolled and randomized
Period: Overall Study
Arm/Group | Active tDCS and Active Exercise | Sham tDCS and Active Exercise | Active tDCS and Sham Exercise | Sham TDCS and Sham Exercise
Started | 28 | 28 | 30 | 30
Completed | 19 | 20 | 20 | 24
Not Completed | 9 | 8 | 10 | 6

BASELINE CHARACTERISTICS:
Population: Baseline participants for randomized subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | Active tDCS and Active Exercise | Sham tDCS and Active Exercise | Active tDCS and Sham Exercise | Sham TDCS and Sham Exercise | Total
Number analyzed (Participants) | 28 | 28 | 30 | 30 | 116
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.8 (12.5) | 46.3 (11.9) | 49.1 (10.2) | 46.2 (13.3) | 47.1 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 24 | 28 | 26 | 103
  Male | 3 | 4 | 2 | 4 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 24 | 23 | 20 | 89
  Not Hispanic or Latino | 5 | 4 | 6 | 6 | 21
  Unknown or Not Reported | 1 | 0 | 1 | 4 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 1 | 1 | 1 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 3 | 3 | 10
  White | 20 | 21 | 23 | 21 | 85
  More than one race | 3 | 3 | 2 | 3 | 11
  Unknown or Not Reported | 1 | 1 | 1 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Conditioning Pain Modulation (CPM)
Description: Pain intensity was measured using the Numeric Pain Scale (NPS; 0 = no pain, 10 = worst pain). Higher scores indicate worse pain. A "pain-6 temperature" was first identified (temperature that elicits NPS = 6).
  Test stimulus: Pain-6 temperature applied for 30s; participants rated pain at 10, 20, and 30s. The test-stimulus score is the average of the three NPS ratings.
  Conditioned stimulus: After 5 minutes, the left hand was immersed in 10-12°C water for 30s while the same pain-6 temperature was applied again. Pain was rated the same way, and the conditioned-stimulus score is the average of the three NPS ratings.
  CPM calculation = (test-stimulus average) - (conditioned-stimulus average). Positive values = better endogenous pain inhibition; negative values = worse.
Time Frame: 6 weeks
Measure: Mean (95% Confidence Interval); unit: Unit on a scale (NPS 0-10)
Arm/Group | Active tDCS and Active Exercise | Sham tDCS and Active Exercise | Active tDCS and Sham Exercise | Sham TDCS and Sham Exercise
Number analyzed (Participants) | 28 | 28 | 30 | 30
Unit on a scale (NPS 0-10) | 0.36 [-0.23 to 0.95] | 0.05 [-0.63 to 0.73] | 0.21 [-0.40 to 0.83] | -0.55 [-1.01 to -0.09]

2. Primary Outcome: Temporal Slow Pain Summation (TSPS)
Description: Participants first determined the temperature that elicited Numeric Pain Scale (NPS) = 6 ("pain-6"). Using this temperature, a train of 15 heat pulses (0.4 Hz) was delivered to the right forearm with a TSA-II thermode.
  Pain was rated using the NPS after the 1st and 15th heat stimulus.
  TSPS calculation:
  TSPS = NPS rating after the 15th stimulus - NPS rating after the 1st stimulus. Higher TSPS values represent greater temporal pain summation (worse outcome).
Time Frame: 6 weeks
Measure: Mean (95% Confidence Interval); unit: Unit on a scale (NPS 0-10)
Arm/Group | Active tDCS and Active Exercise | Sham tDCS and Active Exercise | Active tDCS and Sham Exercise | Sham TDCS and Sham Exercise
Number analyzed (Participants) | 28 | 28 | 30 | 30
Unit on a scale (NPS 0-10) | -0.11 [-0.60 to 0.38] | 0.48 [-0.29 to 1.25] | 0.47 [-0.27 to 1.20] | 0.09 [-0.44 to 0.61]

ADVERSE EVENTS:
Time Frame: 4.5 months
Description: Adverse effects were collected with a questionnaire for adverse effects
Arm/Group | Active tDCS and Active Exercise | Sham tDCS and Active Exercise | Active tDCS and Sham Exercise | Sham TDCS and Sham Exercise
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28 | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28 | 0/30 | 1/30
Other Adverse Events (participants affected / at risk) | 23/28 | 21/28 | 18/30 | 28/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active tDCS and Active Exercise (N=28) | Sham tDCS and Active Exercise (N=28) | Active tDCS and Sham Exercise (N=30) | Sham TDCS and Sham Exercise (N=30)
Allergic reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — The clinicians who treated her reported that the allergic reaction was associated with a poisonous plant around her neighborhood. This adverse event was considered serious as she was admitted for investigation. This event was unrelated.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active tDCS and Active Exercise (N=28) | Sham tDCS and Active Exercise (N=28) | Active tDCS and Sham Exercise (N=30) | Sham TDCS and Sham Exercise (N=30)
Mild Tingling (Skin and subcutaneous tissue disorders) | 23 | 21 | 18 | 28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-13): https://cdn.clinicaltrials.gov/large-docs/25/NCT03371225/Prot_SAP_000.pdf